CLINICAL TRIAL: NCT05884697
Title: Let's K-Talk: A Storytelling Intervention Leveraging Chatbot Technology to Prevent HPV and HPV Associated Cancers for Ethnic Koreans Living in the U.S.
Brief Title: Let's K-Talk - HPV Study for Ethnic Koreans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Minjin Kim, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPV Study for Ethnic Koreans
Record Dates: First submitted 2023-04-03; First posted 2023-06-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Human Papillomavirus Viruses; Papillomavirus Vaccines
Keywords: Korean immigrants; HPV Vaccines; Storytelling Intervention; Korean Americans; Artificial Intelligence Chatbot

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four experimental conditions using a 2x2 factorial design with two factors (Storytelling and Chatbot) and two levels (Yes/On and No/Off). Acceptability and feasibility outcomes include recruitment/retention rates, obtaining photographic documentation, and perceived satisfaction with the intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Qualtrics is an online survey software used by researchers. It can randomly assign participants to different groups without revealing the assignments to participants or researchers, blinding them to the assignment. This ensures unbiased treatment and assessment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- K-Talk Intervention: Storytelling and AI Chatbot (Experimental): After completing the pre-test survey, participants from all intervention groups will receive the written information. Subsequently, they will be randomly assigned to one of the intervention groups. The K-Talk group will receive a series of weekly storytelling videos, and access to the chatbot via the web-based platform KakaoTalk for 3 months.
  Interventions: Other: K-Talk Intervention (Storytelling and K-Bot); Other: Written Information
- Storytelling Intervention (Experimental): After completing the pre-test survey, participants from all intervention groups will receive the written information. Subsequently, they will be randomly assigned to one of the intervention groups. The storytelling intervention group will only be exposed to periodic release of stories via email for 3 months.
  Interventions: Other: Storytelling Intervention; Other: Written Information
- K-Bot (AI Chatbot Intervention) Intervention (Experimental): After completing the pre-test survey, participants from all intervention groups will receive the written information. Subsequently, they will be randomly assigned to one of the intervention groups. The K-Bot group will only interact with the chatbot via the web-based platform or KakaoTalk for 3 months.
  Interventions: Other: K-Bot Intervention; Other: Written Information
- Written Information (Active Comparator): This group will only be exposed to written, didactic HPV education materials after the pre-test.
  Interventions: Other: Written Information

INTERVENTIONS:
Other: K-Talk Intervention (Storytelling and K-Bot) — The K-Talk intervention group receives a combination of a storytelling intervention and an artificial intelligence chatbot (K-Bot) education.
  Arms: K-Talk Intervention: Storytelling and AI Chatbot
Other: Storytelling Intervention — The storytelling intervention features 12 authentic stories from young Korean immigrants and Americans. Each video is about 3 minutes long and includes stories from 1st, 1.5, and 2nd generation young Korean individuals, highlighting their perceptions of HPV and HPV vaccines, and their experiences with HPV vaccination.
  Arms: Storytelling Intervention
Other: K-Bot Intervention — The K-Bot intervention is a conversational and button-based artificial intelligence Chatbot that is available in both English and Korean.
  Arms: K-Bot (AI Chatbot Intervention) Intervention
Other: Written Information — The written information provided includes the Centers for Disease Control and Prevention's (CDC) details on HPV and HPV vaccines.

SUMMARY:
The goal of this clinical trial is to test the feasibility, acceptability, and preliminary efficacy of a storytelling video-based intervention using AI chatbot technology (K-Talk) to promote HPV vaccination behavior among Korean Americans aged 18 to 45.

The main questions this study aims to answer are:

* Is the K-Talk intervention feasible for use among Korean Americans aged 18 to 45?
* Is the K-Talk intervention acceptable to the target population?
* What is the preliminary efficacy of the K-Talk intervention in promoting HPV vaccination uptake?

Participants will be Korean Americans aged 18 to 45 who are at risk for HPV infection. Participants will be asked to complete a baseline survey and then will be "randomized" into one of four groups: Group 1 (chatbot + storytelling intervention), Group 2 (chatbot only), Group 3 (storytelling only), and Group 4 will be only exposed to written didactic HPV education materials. All groups will receive written didactic HPV education materials. Researchers will compare how Group 1, a combination of AI Chatbot and storytelling intervention is more effective than other intervention groups in promoting HPV vaccination uptake among underserved, hard-to-reach Korean Americans.

DETAILED DESCRIPTION:
The objective of this study is to conduct a pilot Multiphase Optimization Strategy trial (MOST) to evaluate the acceptability, feasibility, and preliminary efficacy of K-Talk as an intervention to improve HPV vaccination initiation and completion among Korean American men and women. K-Talk is a user-centered intervention that combines AI chatbot technology with storytelling to enhance health communication, foster connection, and provide accurate advice related to HPV vaccination. The study design follows an optimization phase of the MOST, utilizing a 2 x 2 factorial design with two factors (storytelling and chatbot) and two levels (Yes/On and No/Off). The study aims to recruit a total of 160 participants, with 40 participants assigned to each experimental condition. The sample will consist of 80 males and 80 females who are eligible for participation in factorial experimentation using the MOST design. Interested individuals will undergo an online eligibility screening survey. If eligible for the study, participants will receive an online survey link containing informed consent, a baseline survey, written HPV information, and random assignment to an intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Identify as a Korean ethnic person
2. Reside in the U.S.
3. between the ages of 18 and 45
4. be able to speak or read English
5. not have been vaccinated against HPV
6. use a mobile device.

Exclusion Criteria:

1. Participants who do not identify as a Korean ethnic person
2. Participants who do not reside in the U.S.
3. Participants who are not between the ages of 18 and 45.
4. Participants who cannot speak or read English.
5. Participants who have been vaccinated against HPV.
6. Participants who do not use a mobile device.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed 3 doses of HPV vaccines at 12-months | 12 months after the baseline
  Completion of 3 doses of HPV vaccines
Number of participants who completed 3 doses of HPV vaccines at 6-months | 6 months after the baseline
  Completion of 3 doses of HPV vaccines
Number of participants who received at least one dose of HPV vaccine at 3-month | 3-months after the baseline
  Participants who received at least one dose of HPV vaccine at 3-month
Number of participants who received at least one dose of HPV vaccine at 6-month | 6-months after the baseline
  Participants who received at least one dose of HPV vaccine at 6-month
Number of participants who received at least one dose of HPV vaccine at 12-month | 12-months after the baseline
  Participants who received at least one dose of HPV vaccine at 12-month

SECONDARY OUTCOMES:
Assessment of Knowledge about HPV and HPV Vaccines: A 34-Item Survey (True/False/I don't know) | at baseline and 3-month follow-up
  Higher scores represent better knowledge.
Assessing Perceived Risk of HPV and Other STIs: A 17-Item Survey (on a 1-5 Likert scale) | at baseline and 3-month follow-up
  Higher scores indicate higher risk perceptions about HPV and STI
Assessment of Intention to Receive HPV Vaccine: Two Items Self-Report | at baseline, 3-month, 6-month, and 12-month follow-up
  Two questions will be used to assess participants' intention to receive HPV vaccines: "Do you intend to get the HPV vaccine?" and "How likely is it that you will get an HPV vaccine in the next 3 months?"

CONTACTS AND LOCATIONS:
Overall Officials: Minjin Kim, PhD., RN, Principal Investigator — UC College of Nursing
Locations (1):
- Minjin Kim, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Sharing only aggregated data will be presented in a summary format without any identifying information about individual participants.